CLINICAL TRIAL: NCT06740604
Title: Evaluation of the Efficacy and Safety of the BSD-10CH Transcranial Direct Current Stimulation Device for Temporary Improvement of Upper Limb Function in Stroke Patients: a Single-Center, Randomized, Blinded, Parallel-Design Investigator-Initiated Clinical Trial
Brief Title: BSD-10CH TDCS for Upper Limb Function Improvement in Stroke Patients: a Randomized Clinical Trial
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Pusan National University Yangsan Hospital (Other)
Responsible Party: Principal Investigator, Yong-il Shin, Professor, Pusan National University Yangsan Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 23-2024-004
Record Dates: First submitted 2024-12-13; First posted 2024-12-18 (Actual); Last update posted 2024-12-18 (Actual); Status verified 2024-12

CONDITIONS: Stroke; TDCS
Keywords: Stroke; tDCS
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- BSD-10CH (Experimental): The BSD-10CH stimulation was applied five times a week for 4 weeks, with each session lasting 20 minutes per day.
  Interventions: Device: BSD-10CH
- Sham BSD-10CH (Sham Comparator): The Sham BSD-10CH stimulation was applied five times a week for 4 weeks, with each session lasting 20 minutes per day.
  Interventions: Device: Sham BSD-10CH

INTERVENTIONS:
Device: BSD-10CH — The BSD-10CH stimulation was applied five times a week for 4 weeks, with each session lasting 20 minutes per day.
  Arms: BSD-10CH
Device: Sham BSD-10CH — The Sham BSD-10CH stimulation was applied five times a week for 4 weeks, with each session lasting 20 minutes per day.
  Arms: Sham BSD-10CH

SUMMARY:
This clinical study compares the effectiveness and safety of the BSD-10CH transcranial direct current stimulation (tDCS) device, applied alongside rehabilitation therapy, with a control device in stroke patients. After 4 weeks of treatment, the study evaluates the transient improvement in motor cortex activation and upper extremity function between the two groups.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 19 years or older.
* Diagnosed with stroke based on clinical observation and neuroimaging.
* First-time stroke patients (1st stroke).
* Stroke onset between 2 weeks and 12 months prior to screening.
* Stroke lesion located in the cortex or subcortex.
* Presence of hemiparesis in the upper limb.
* Upper limb FMA score of 53 or lower.
* Ability to read and understand the informed consent form, and to respond to questionnaires.
* Willing to voluntarily participate in the clinical trial, and able to provide written informed consent to participate throughout the study period.

Exclusion Criteria:

* Recurrent stroke, traumatic brain injury, spinal cord injury, degenerative neurological diseases (such as Parkinson's disease), or other conditions affecting upper limb function.
* MMSE score of 19 or lower, indicating dementia, and inability to follow study instructions.
* Global aphasia or communication disorders.
* Brain injury caused by trauma, ischemia, hypoxia, or similar conditions.
* Uncontrolled medical or surgical conditions.
* Skin inflammation or other dermatological issues that may prevent attachment of tDCS electrodes.
* Medical contraindications for the use of tDCS devices (e.g., pacemaker, aneurysm clips, prosthetic heart valves, cochlear implants, or other implanted metal devices).
* Previous use of similar stimulation devices or participation in related clinical trials within the last year.
* History of major psychiatric disorders (e.g., major depressive disorder, schizophrenia, bipolar disorder, or dementia) within the past 5 years.
* History of epilepsy (seizures) within the past 5 years.
* History of substance abuse (e.g., neuroleptics, sedatives, narcotics, or illicit drugs) within the past 5 years.
* Participants requiring changes in medications that could affect cognitive or motor function during the study (unless the participant has been on stable, prohibited medications for at least 3 months).
* History of alcohol addiction treatment within the last 5 years.
* Severe visual impairment that cannot be corrected with glasses, preventing the reading of standard print.
* Hearing impairment that prevents communication, even with hearing aids.
* Difficulty breathing at rest.
* A history of suicide attempts within the past 6 months.
* Pregnant or breastfeeding women, or men and women of reproductive age who do not agree to use appropriate contraception throughout the study. *Acceptable methods of contraception include:

  * Hormonal methods (oral contraceptives, injections, patches, implants, etc.)
  * Surgical sterilization (vasectomy, bilateral tubal ligation)
  * Dual protection (male condoms, diaphragm, cervical cap)
  * Intrauterine devices or systems.
* Pregnant or breastfeeding participants.
* Any other clinical condition deemed by the investigator to make the participant unsuitable for the study.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2024-02-21 (Actual); Primary Completion 2024-08-01 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in Oxy-Hemoglobin Concentration Description | Baseline and Week 4(Visit 22)
  Functional Near-Infrared Spectroscopy (fNIRS) will be used to measure changes in oxy-hemoglobin concentration in the brain, reflecting alterations in cerebral blood flow and neurovascular reactivity (NVR) during transcranial direct current stimulation (tDCS). fNIRS works by detecting changes in the absorption, scattering, and reflection of near-infrared light (ranging from 800 nm to 2500 nm), which are associated with the concentration changes of oxy-hemoglobin and deoxy-hemoglobin. This technique allows for the assessment of cerebral oxygenation, blood flow, and energy metabolism, providing insights into neurovascular coupling.
Change in Upper Extremity Function Score of the Korean Version of the Fugl-Meyer Assessment (K-FMA) | Baseline and Week 4(Visit 22)
  The Korean version of the Fugl-Meyer Assessment (K-FMA) is a tool used to evaluate the recovery of upper extremity function in stroke patients with hemiplegia. It assesses sensory and motor function through 63 items, with a total score ranging from 0 to 126 points. The assessment covers categories such as shoulder, elbow, forearm, wrist, hand, upper extremity coordination, sensation, passive joint movement, and joint pain during passive movement. Recovery is measured by comparing the baseline score to the score after 4 weeks.
Change in Grip and Pinch Strength | Baseline and Week 4(Visit 22)
  Grip strength is measured using the Jamar Hydraulic Hand Dynamometer (5030J1). The handle is fixed at level II regardless of hand size. Pinch strength is measured using the Jamar Pinch Gauge (PG 60). First, grip strength is measured on both sides, followed by the measurement of tip pinch strength on both sides. Subsequently, 3-jaw pinch and lateral pinch strengths are measured in the same manner. After a 5-minute rest, grip strength and the three types of pinch strengths are measured again to calculate the average. Tip pinch measures the force between the thumb and index finger tip, lateral pinch measures the force between the thumb and the side of the index finger, and 3-jaw pinch measures the force between the thumb and the index-middle finger. During grip strength measurement, the subject sits in a chair with the shoulder adducted and not rotated, the elbow flexed at 90°, and the forearm and wrist in a neutral position. The scores are recorded in grams (g).
Change in Korean-Modified Barthel Index (K-MBI) score | Baseline and Week 4(Visit 22)
  The K-MBI is an assessment tool used to evaluate a patient's ability to perform activities of daily living. It consists of 10 items that measure the level of independence or dependence in tasks such as personal hygiene, bathing, eating, toileting, mobility, stair climbing, dressing, bowel and bladder control, transfers between chair/bed, and using a bathtub or shower. Scores range from 0 (completely dependent) to 100 (completely independent). The change is calculated by subtracting the baseline score from the Week 4 score.

CONTACTS AND LOCATIONS:
Overall Officials: Young-Il Shin, Dr., Study Director — Pusan National University Yangsan Hospital
Locations (1):
- Pusan national university Yangsan Hospital, Gyeongsang, Yangsan, South Korea

IPD SHARING:
Plan to Share IPD: No